CLINICAL TRIAL: NCT05538234
Title: Biomarkers of Kidney Function in Transplant Medicine
Status: Recruiting | Type: Observational
Sponsor: University Hospital Ostrava (Other)
Responsible Party: Sponsor
Other Study IDs: KARIM-827/2021
Record Dates: First submitted 2022-09-09; First posted 2022-09-13 (Actual); Last update posted 2023-09-07 (Actual); Status verified 2023-09

CONDITIONS: Acute Kidney Injury
Keywords: organ donor; organ recipient; transplant medicine; acute kidney injury
MeSH Terms: conditions — Acute Kidney Injury | interventions — Transplantation; Tissue and Organ Harvesting; Organ Transplantation

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Blood samples will be collected from the study participants.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Non-living organ donors: Group of non-living donors
  Interventions: Diagnostic Test: Laboratory values - baseline; Other: Medical information 12 hours before organ harvesting; Other: Medical information during organ harvesting/transplantation; Procedure: Organ harvesting
- Living organ donors: Group of living organ donors
  Interventions: Diagnostic Test: Laboratory values - baseline; Diagnostic Test: Laboratory values - 12 hours after reperfusion; Diagnostic Test: Laboratory values - 48 hours after reperfusion; Diagnostic Test: Laboratory values - 7 days after reperfusion; Diagnostic Test: Laboratory values - 90 days after reperfusion; Other: Medical information during organ harvesting/transplantation; Procedure: Organ harvesting
- Organ recipients: Group of organ recipients
  Interventions: Diagnostic Test: Laboratory values - baseline; Diagnostic Test: Laboratory values - 12 hours after reperfusion; Diagnostic Test: Laboratory values - 48 hours after reperfusion; Diagnostic Test: Laboratory values - 7 days after reperfusion; Diagnostic Test: Laboratory values - 90 days after reperfusion; Other: Medical information during organ harvesting/transplantation; Procedure: Organ transplantation

INTERVENTIONS:
Diagnostic Test: Laboratory values - baseline — Baseline laboratory values will be obtained
Other: Medical information 12 hours before organ harvesting — * average hourly diuresis
  * hypotension MAP<65 Torr longer than 30 minutes (YES/NO)
  * Furosemide administration (YES/NO)
  * Mannitol administration (YES/NO)
  * administration of anti-diuretic hormone (YES/NO)
  * administration of vasopressors (YES/NO)
  * polyuria >3ml/kg/h (YES/NO)
  * nephrotoxic agents during hospitalization (YES/NO)
  Groups: Non-living organ donors
Diagnostic Test: Laboratory values - 12 hours after reperfusion — Laboratory values will be obtained 12 hours after reperfusion
  Groups: Living organ donors; Organ recipients
Diagnostic Test: Laboratory values - 48 hours after reperfusion — Laboratory values will be obtained 48 hours after reperfusion
  Groups: Living organ donors; Organ recipients
Diagnostic Test: Laboratory values - 7 days after reperfusion — Laboratory values will be obtained 7 days after reperfusion
  Groups: Living organ donors; Organ recipients
Diagnostic Test: Laboratory values - 90 days after reperfusion — Laboratory values will be obtained 90 days after reperfusion
  Groups: Living organ donors; Organ recipients
Other: Medical information during organ harvesting/transplantation — Medical information during organ harvesting/transplantation
  * hypotension MAP 65 Torr > 5 minutes (YES/NO)
  * vasopressor support (YES/NO, duration in minutes)
Procedure: Organ harvesting — Organ harvesting for transplant
  Groups: Living organ donors; Non-living organ donors
Procedure: Organ transplantation — Transplantation of the harvested organ
  Groups: Organ recipients

SUMMARY:
Biomarkers of kidney function in transplant medicine is an international, multicentre, observational, non-interventional study.

The project is aimed at monitoring biomarkers of acute kidney dysfunction in deceased organ donors, living organ donors, and organ recipients.

DETAILED DESCRIPTION:
The study is observational, without any changes from the standard care, including only selected laboratory assessments, from standard blood samples collected from the donors/recipients.

Informed consent will be required from living donors and recipients.

The mainly used current criteria of organ acceptability in transplant medicine include urine output and laboratory parameters of acute kidney dysfunction - serum levels of urea and creatinine. Literary sources show that these classic criteria of kidney dysfunction develop only with a significant reduction of (glomerular and tubular) kidney functions and return to normal only slowly after the function of the kidneys has been restored.

New possibilities of early kidney dysfunction diagnostics are being studied, using more sensitive tests - determination of biomarkers of acute kidney dysfunction. These may serve as decisive criteria for the safe use of organs from so-called marginal donors and identify early serious impairment of kidney function in donors with preserved urine output, without fulfilled criteria of acute kidney injury.

ELIGIBILITY:
Inclusion Criteria:

* age 18+
* signed Informed Consent in case of living organ donors and recipients
* fulfillment of all legal requirements for organ harvesting from a deceased donor
* fulfillment of all ethical principles of end-of-life patient care
* medical suitability of organs for transplant use

Exclusion Criteria:

- disapproval of family members with the enrolment of the patient in the study

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Living and deceased organ donors, organ recipients.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2023-01-01 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-03-31 (Estimated)

PRIMARY OUTCOMES:
Sensitivity of kidney dysfunction biomarkers | up to 90 days after the procedure
  Sensitivity of kidney dysfunction biomarkers will be assessed using the Kidney Donor Risk Index and Kidney Donor Profile Index

SECONDARY OUTCOMES:
Comparison of levels of kidney dysfunction biomarkers between DBD donors (Donation after Brain Death) and DCD donors (Donation after Cardiac Death | during baseline data collection
  levels of kidney dysfunction biomarkers between DBD donors (Donation after Brain Death) and DCD donors (Donation after Cardiac Death will be assessed.
Correlation of Acute Kidney Injury biomarkers in DCD donors with the time of warm ischemia | during organ harvesting
  Correlation of Acute Kidney Injury biomarkers in DCD donors with the time of warm ischemia will be assessed.
Predictive value of Acute Kidney Injury biomarkers in organ recipients | up to 90 days after transplantation
  The predictive value of Acute Kidney Injury biomarkers in organ recipients for worsened function of the transplanted kidney will be assessed
Association between donor kidney dysfunction with selected risk factors | up to 90 days after transplantation
  Association between donor kidney dysfunction with selected risk factors will be assessed (ion disbalance, circulatory instability)

CONTACTS AND LOCATIONS:
Overall Officials: Peter Sklienka, MD, Ph.D., Principal Investigator — University Hospital Ostrava
Locations (1):
- University Hospital Ostrava, Ostrava, Moravian-Silesian Region, Czechia

IPD SHARING:
Plan to Share IPD: No
Individual participant data may be provided upon request.